CLINICAL TRIAL: NCT07104058
Title: A Prospective Study on the Effect of Minimal Residual Disease Detected by Fibroblast Activation Protein PET / CT on the Recurrence of IgG4-related Disease
Brief Title: A Study on the Effect of MRD Detected by FAPI PET / CT on the Recurrence of IgG4-RD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luo Yaping (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Luo Yaping, Medical Doctor (M.D.), Chief Physician, Professor, Assistant Director, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-IgG4RD; Categoty C, UBJ10707 (Other Grant/Funding Number: PekingUMCH Talent Cultivation Program)
Record Dates: First submitted 2025-05-07; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: IgG4-Related Diseases
Keywords: IgG4-Related Diseases; FAPI PET/CT
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(68Ga-FAPI PET / CT negative patients) (Other): Group A (MRD-negative) will receive no intervention and enter treatment withdrawal with observational follow-up.
  Interventions: Diagnostic Test: 68Ga-FAPI PET / CT
- B(68Ga-FAPI PET / CT positive patients) (Other): Group B (68Ga-FAPI PET/CT positive, indicating MRD-positive status). Group B (MRD-positive) patients will be randomized 1:1 into either the experimental subgroup B1 (continuing low-dose glucocorticoids with or without immunosuppressant maintenance therapy) or the control subgroup B2 (treatment withdrawal with observational follow-up).
  Interventions: Diagnostic Test: 68Ga-FAPI PET / CT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI PET / CT — IgG4-RD patients with clinical complete remission after hormone and immunosuppressive therapy and 18F-FDG PET / CT negative were included. After enrollment, 68Ga-FAPI PET / CT screening was performed.

SUMMARY:
This study intends to use the new technology of fibroblast activation protein PET / CT to study whether the tiny residual lesions detected by 68Ga-FAPI PET / CT are related to the recurrence of IgG4-RD in patients with IgG4-RD who have been clinically evaluated for complete remission after treatment.

DETAILED DESCRIPTION:
This prospective randomized controlled study will enroll IgG4-RD patients who have achieved clinical complete remission with negative 18F-FDG PET/CT findings after glucocorticoid and immunosuppressant therapy. Following enrollment, all participants will undergo 68Ga-FAPI PET/CT screening.Based on the results, patients will be stratified into two groups: Group A (68Ga-FAPI PET/CT negative, indicating MRD-negative status) and Group B (68Ga-FAPI PET/CT positive, indicating MRD-positive status). Group A (MRD-negative) will receive no intervention and enter treatment withdrawal with observational follow-up. Group B (MRD-positive) patients will be randomized 1:1 into either the experimental subgroup B1 (continuing low-dose glucocorticoids with or without immunosuppressant maintenance therapy) or the control subgroup B2 (treatment withdrawal with observational follow-up). All participants will be followed for 18 months with quarterly clinical disease activity assessments to document relapse. Randomization will be performed using an online randomization system, with only the endpoint assessors blinded to group allocation while other investigators and study subjects remain aware of the randomization results.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years old ;
2. Meet the 2019 ACR / EURLAR IgG4-RD diagnostic criteria ;
3. The disease was stable for more than 1 year, and the clinical evaluation of the disease was complete remission * ;
4. Glucocorticoid dosage ≤ prednisone 7.5mg / d × 6 months or more, or combined with an immunosuppressive therapy ( mycophenolate mofetil ) Ester ≤ 1.0g / d, leflunomide ≤ 20mg / d, methotrexate ≤ 15mg / w, azathioprine ≤ 100mg / d, iguratimod ≤ 25mg Bid )

Exclusion Criteria:

( 1 ) Combined with other connective tissue disease patients ( 2 ) patients with tumor ; ( 3 ) women during pregnancy or planning pregnancy ; ( 4 ) active infection, including HIV, HCV, HBV, TB, etc. ; ( 5 ) Severe irreversible organ damage ; ( 6 ) In the active stage of the disease, the IgG4-RD reaction index score of the single affected organ was 2 points ; ( 7 ) stable condition less than 1 year ; ( 8 ) patients who relapsed within 1 year of previous hormone reduction and withdrawal ; ( 9 ) Combination of two or more immunosuppressive agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of IgG4-related disease. | 18 months after enrollment
  All participants will be followed for 18 months with quarterly clinical disease activity assessments to document relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Yaping LUO, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No